CLINICAL TRIAL: NCT05840120
Title: PTSD Clinical Trials Review: Examining Patient Experiences in PTSD Clinical Trials to Identify Influencing Factors
Brief Title: Studying the Clinical Research Experiences of Patients With PTSD
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 80684805
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: PTSD
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical research participation percentages haven't always been fully representative of a given demographic.

The goal is to find out which aspects of a clinical study may make it more difficult for patients to take part or see it through.

The data will be evaluated through different demographic lenses and identify trends that could help improve the experience of future PTSD patients during clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Must have a medical diagnosis of PTSD that has been confirmed by a physician.
* Aged ≥ 18 years old and ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed.
* Willing and able to comply with scheduled visits, treatment schedule, laboratory tests and other requirements of the study.

Exclusion Criteria:

* Pregnant or lactating woman
* Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent.
* Known medical condition that, in the investigator's opinion, would increase the risk associated with study participation or study drug(s) administration or interfere with the interpretation of safety results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PTSD patients who are actively considering involvement in an observational clinical trial, but have not yet completed enrollment and registration.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a PTSD medical study. | 3 months
Number of PTSD patients who remain in clinical trial until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ronconi JM, Shiner B, Watts BV. Inclusion and exclusion criteria in randomized controlled trials of psychotherapy for PTSD. J Psychiatr Pract. 2014 Jan;20(1):25-37. doi: 10.1097/01.pra.0000442936.23457.5b. PMID 24419308
- [Background] Sofuoglu M, Rosenheck R, Petrakis I. Pharmacological treatment of comorbid PTSD and substance use disorder: recent progress. Addict Behav. 2014 Feb;39(2):428-33. doi: 10.1016/j.addbeh.2013.08.014. Epub 2013 Aug 22. PMID 24035645
- [Background] Steenkamp MM, Litz BT, Hoge CW, Marmar CR. Psychotherapy for Military-Related PTSD: A Review of Randomized Clinical Trials. JAMA. 2015 Aug 4;314(5):489-500. doi: 10.1001/jama.2015.8370. PMID 26241600

DOCUMENTS (1):
  • Informed Consent Form (2023-04-21): https://cdn.clinicaltrials.gov/large-docs/20/NCT05840120/ICF_000.pdf